CLINICAL TRIAL: NCT03057340
Title: The Treatment of Advanced Lung Cancer With Dribbles Antigen by Targeting
Brief Title: The Treatment of Advanced Lung Cancer With Dribbles Antigen by Targeting Activation of Tcells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pl001
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Advanced non-small cell lung cancer; Dribbles
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sialorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DRibble vaccine (Experimental): Blood samples collection: collect of 10ml patients peripheral blood, separate PBMC;Day 1: DRibble group guided by ultrasound in patients with inguinal lymph nodes injected the DRibble vaccine;Day8: collecte 50 ml peripheral blood and separate monocytes and lymphocytes;Intensify immune cells amplification;Identification of immune cell;Detection of Immune cells microbial;20-22 days: immune cells back to patients;55 days: collecte 10 ml peripheral blood, after the separation of PBMC in vitro induced to DC, cocultivate with DRibble and subcutaneous injection at 60th day;Day 75: collecte 10 ml peripheral blood, separate PBMC and detecte T cell immune response ability.
  Interventions: Biological: Dribble vaccine

INTERVENTIONS:
Biological: Dribble vaccine — DRibble vaccine with DC/CIK(The experimental group) DRibble vaccine will be administered at day1,22,55

SUMMARY:
Malignant tumor has become the leading cause of death in humans, and the number one killer in malignant tumor is the lung cancer. Intensifying environmental pollution comes with rising of the incidence of lung cancer and the high mortality,what's the worst that the 5-year survival rate is only about 15%, accounting for first place in the malignant tumors, Exploiting for novel antitumor technology and products comes to arrest growing attention of the governments and businesses because of the uneffectively curbing of tumor threat to people's life and health on conventional three treatments (surgery, radiotherapy and chemotherapy). Biological and immunotherapy was voted to one of the ten big breakthrough in 2013 by Science magazine, and considered as a new development direction for cancer treatment in the 21st century.

The existing immune treatment mainly includes: adoptive immune therapy, tumor vaccine therapy, immune checkpoint-antibody therapy and other auxiliary therapy, and the adoptive immunotherapy was researched and developeded former in addition the most mature treatment among these therapies.

Recently, Dr Hu Hong - Ming's team put forward an innovative cancer treatment strategy: using of autophagy role to capture tumor antigen for preparation of tumor vaccine. In this strategy, the blocking proteasome activity of in vitro cultured tumor cells dealed with Bortezomib (proteasome inhibitors) causes enrichment of short-lived protein (SLiPs) and misfolded proteins (DRiPs) in autophagosome,called DRibbles corpuscle. Tumor vaccine maded from collecting these DRibbles corpuscle preparation as, also known as the DRibble vaccine.

At present, clinical research has been carried out about Dribble liver cancer vaccine unit with DC - CIK therapy in liver cancer in the second hospital of Nanjing nearly four years,and more than 300 cases has been completed. Clinical research results show that Dribble vaccine has good security, producing stronger immune response compared with the DC-CIK therapy alone. But it is still no cognization for the efficacy and safety of DC-CIK joint DRibble lung cancer vaccine in China, whether it is better than the current DC - CIK immune therapy, needed for further clinical research and expected to provide a better immune treatment for NSCLC patients.

DETAILED DESCRIPTION:
Malignant tumor has become the leading cause of death in humans, and the number one killer in malignant tumor is the lung cancer. Intensifying environmental pollution comes with rising of the incidence of lung cancer and the high mortality,what's the worst that the 5-year survival rate is only about 15%, accounting for first place in the malignant tumors, Exploiting for novel antitumor technology and products comes to arrest growing attention of the governments and businesses because of the uneffectively curbing of tumor threat to people's life and health on conventional three treatments (surgery, radiotherapy and chemotherapy). Biological and immunotherapy was voted to one of the ten big breakthrough in 2013 by Science magazine, and considered as a new development direction for cancer treatment in the 21st century.

The existing immune treatment mainly includes: adoptive immune therapy, tumor vaccine therapy, immune checkpoint-antibody therapy and other auxiliary therapy, and the adoptive immunotherapy was researched and developeded former in addition the most mature treatment among these therapies. The adoptive immunotherapy has been carried out in many units primarily is the autologous DC - CIK immunotherapy,which called the Dendritic cells (Dendritic cells, DC) and Cytokine Induced Killer cells (Cytokine Induced Killer, CIK) immunotherapy. The principle of this technology is: separating of monocytes and lymphocytes of human peripheral blood, then ugmentated and activated by a variety of cytokines in vitro (e.g., IFN - gamma, IL - 1, IL - 2, anti - CD3 mAb) to a mixed lymphocyte with antigen presenting and broad-spectrum function of killing tumor cells. The amplifying activated DC-CIK intravenous back to patients, releasing of active substances such as CIK cells perforin,and grain enzyme B to tumor cells after combining with the tumor cells in the body, which dissolves the tumor cells.Meanwhile the secreting of a variety of cytokines, such as IL - 2, IFN - gamma and TNF alpha, improves the body's immune function, and gives the role of anti-tumor function.

Existing literature report and our previous study in biological treatment center showed that good safety, small side effects and good tolerance for the vast majority of patients. In curative effect, the current report reveals DC-CIK technology has a good curative effect maidly on leukemia, lymphoma, ovarian cancer, stomach cancer, etc., except for lung cancer.It could because of the complex lung cancer tumor antigen,or weak tumor specific T cell response. How to improve the effectiveness of the presented lung cancer antigen and stimulate stronger tumor specific T cell response needs to be addressed in improving the curative effect of the lung cancer immunotherapy.

In recent years checkpoint point antibody therapy has a breakthrough in tumor immunotherapy, including CTLA-4, PD - 1 and PD - L1. a number of clinical studies revealed the therapy of PD - 1 and PD - L1 antibody for advanced NSCLC, especially in lung squamous carcinoma has good treatment effect, and the disease objective response rate achieve 10-23%. Autologous DC/CIK therapy has been widely carried out in domestic,and has a good security proved by many clinical practice.As the lack of effective tumor antigen, there are no large randomized, double-blind study confirm its function in extending patient survival and preventing tumor progression so far. Some hospitals adopted the tumor cell lysis solution or single molecule protein peptide/DC united CIK technology, which means to load tumor cell lysis or single molecule protein peptide as a tumor antigen to DC unite with in vitro induced CIK at the same time.When compared to CIK therapy alone, the unit therapy can not only non-specificly damage tumor,but also induce the body to produce tumor-specific immune response.However most of the tumor antigens contained in tumor cell lysis are longevity protein that cannot be effectively intaken by DC,leading to limited effective antigen presented by DC to T lymphocyte. In addition, the tumor antigen longevity protein can exist for a long time in the natural growth of tumor cells, and can be recognized by the patients for its own organization,therefore immune tolerance inhibites the immune response affecting the effect of killing tumor. Single molecule protein polypeptide only induce specific immune response to a single or a few tumor antigen, not the mutatd tumor antigen,resulting in escape of tumor. We need to develop new cell treatments because of autologous DC/CIK therapy can not produce effective immune response ,for providing a new aiternative candidate to unite checkpoint antibody therapy in the future.

Recently, Dr Hu Hong - Ming's team put forward an innovative cancer treatment strategy: using of autophagy role to capture tumor antigen for preparation of tumor vaccine. In this strategy, the blocking proteasome activity of in vitro cultured tumor cells dealed with Bortezomib (proteasome inhibitors) causes enrichment of short-lived protein (SLiPs) and misfolded proteins (DRiPs) in autophagosome,called DRibbles corpuscle. Tumor vaccine maded from collecting these DRibbles corpuscle preparation as, also known as the DRibble vaccine.Our early studies have suggested that the DRibble tumor vaccines are more powerful than the tumor cell vaccine, because the whole tumor cell vaccine does not contain easily degradated short-lived proteins which cannot be cross presented to DC efficiently. These short-lived protein avoid being degradated by the proteasome in the DRibble vaccine, and packaged into autophagosome vesicles with double membrane structure. These vesicles contain endogenous risk signaling molecules (such as HSP90, HMGB1, etc.), can effectively trigger the congenital immune response. Therefore, when co-culture with once DRibble vaccine,DC can effectively intake DRibble vaccine and presenting tumor related antigen to the DC surface, combining with MHC molecules to activate T cells, resulting in the immune response. Compared with whole lung cancer vaccine, DRibble lung cancer vaccines can provide a wider range of tumor associated antigen, make the body no longer keep the tolerance for lack of cross presented, which can cause strong immune response. Dr Hu Hong Ming's team have also found that allogeneic Dribble can induce equally effective immune response compare with autologous tumor cells DRibble vaccine and tumor regression, the result has been confirmed in multiple tumor models. Due to the lack of classic MHC molecules,DRibble vaccine proteins can be rapidly degradated by DC, and allogeneic DRibble vaccine would not induce adverse effects due to the induction of allograft immune response, remaindering it's safety and efficacy.

DRibble surface have a large number of target molecular ligands of DC,directely combine with xDC cells with high expression CLEC9A on surface. xDC cells can efficiently cross presente antigen to DC, thus can improve the efficiency of presenting DRibble antigen. Besides, immune response induce by DRibble have immune memory and identify a wide variety of tumor specific antigen, it will amplificate palying against tumor cells regeneration and prevent tumor escape when stimulated again.By Providence cancer centers in the United States for nearly 10 years of research, the safety of the DRibble has been fully validated by Ⅰ/Ⅱ clinical trials.

Based on the above research foundation, our project intends to carry out the following research: 1. The curative effect and the influence of the overall survival of late-stage NSCLC patients after receivie new DRibble vaccine, and compared with the existing DC/CIK therapy efficacy, 2. Further study the mechanism of Dribble vaccine therapy effects on human lung cancer cells, system analysis and evaluate the clinical curative effect and promotion value.

Research objects: this study intends to include ⅢA/ⅢB/Ⅳ period non-small cell lung cancer without radical prostatectomy (about 60% of the total number), patients who received 2-6 courses of chemotherapy, accept or not accept radiation therapy and disease control stage. Selected patients were randomly divided into new immunotherapy and conventional DC/CIK treatment group.

Therapeutic schedule: This trial of allogeneic DRibble vaccine unite with DC/CIK or DC/CIK alone for Treatment of Stage IIIA or B NSCLC. Two arms will be studied. 30 patients will be randomized to arm 1 and 2.

Arm1: DRibble vaccine with DC/CIK(The experimental group) Arm2: DC/CIK(The control group) Methods and procedures

1. Hospital ethics committee approval.
2. Recruting the appropriate patients according to the inclusion criteria and exclusion criteria .
3. Sign the patients informed consent
4. The preparation of DRibble lung cancer vaccines
5. Blood samples collection: collecte of 10ml patients peripheral blood, separate PBMC as before treatment reference specimens.
6. Day 1: DRibble group guided by ultrasound in patients with inguinal lymph nodes under the vaccine of inject DRibble, the control group no injections
7. Day8: collecte 50 ml peripheral blood and separate monocytes and lymphocytes
8. Intensify immune cells amplification (biological treatment center) : using CD3 antibodies activation, IL - 2 promotes lymphocytes proliferation for the killing cells;GM-CSF induce mononuclear cells differentiation for DC, joint immune treatment group to DRibble vaccine co-culture with DC cells for 24h in Dribble unit with DC/CIK group.
9. Identification of immune cell (clinical laboratory, biological treatment center) : counting cell number, cell activity, the surface markers.
10. Detection of Immune cells microbial (clinical laboratory, biological treatment center) : bacteria, mycoplasma and endotoxin.
11. 20-22 days: immune cells back to patients: physiological saline washing cells, venous return after suspension, within a period of treatment by several times.
12. 55 days: collecte 10 ml peripheral blood, after the separation of PBMC in vitro induced to DC, cocultivate with DRibble and subcutaneous injection at 60th day.
13. Day 75: collecte 10 ml peripheral blood, separate PBMC and detecte T cell immune response ability.

System evaluation the therapeutic effect and promotion value of Dribble: 1.The clinical evaluation of curative effect: comparing the experimental group and control group of progression-free survival and overall survival, drawing survival curve, and statistically analyzed. 2. evaluating DRibble immune response , comparing the first time collected peripheral blood with the treated peripheral blood and follow-up stage, immune function detected of testing mainly included below: in vitro testing level of DRibble specific T cells in the peripheral blood before and after the treatment, in order to make clear the antigen produced specific immune response; culturing the specific T cells in vitro,carrying out recognition experiment and patients autologous tumor (if successful separated) and multiple builded strains lung cancer cells isolated from patients in vitro, in order to make clear the specific T cells generated by experimental group could recognize many strains of lung cancer cells, means allogeneic DRibble specific T cells can response to different patient's tumor cells. 3. Safety evaluation indexes: adverse reaction(Redness and swelling, pain, skin rashes, itching, etc. Allergic reactions);The blood test index is in accordance with the standard(Routine blood, liver and kidney function, electrolyte, etc);The quality of life (Weight and BMI, blood protein level, physical strength grade, psychological, emotional evaluation, etc).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years old, pathological diagnosis of advanced non-small cell lung cancer, after treatment with radiation and chemotherapy and (or) targeted drugs disease still progress.
* Clear that heart, lung, liver, kidney at physical basic normal, and basic normal immune system function.
* No allergic reaction of biological products, asthma and other allergic constitution.
* A patient or his legal representative signed informed consent.

Exclusion Criteria:

* The obvious blood coagulation dysfunction patients.
* Patients infected with tuberculosis, hepatitis b, AIDS and syphilis positive diseases.
* Severe diabetes, high blood pressure, stroke, heart failure, and kidney disease.
* Autoimmune diseases such as systemic lupus erythematosus (sle) and Rheumatoid arthritis (ra)
* Large doses or long-term glucocorticoid, and other immunosuppressive users (more than 4 weeks).
* Pregnant and nursing women has a history of allergies of biological products.
* Collect blood and doping in another place.
* Allergies or active infection that effect the observation of Tolerance activity.
* Heart, lung, liver, kidney or bone marrow function obviously low.
* Unable or unwilling to sign a consent form or to comply with the technical requirement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Evaluate progression-free survival. Tumor measurements by CT scan will be obtained at week 16 and subsequently at the discretion of the treating investigator. After the treatment period, patients will be seen every 3 months for 2 years, or until progressive disease.

SECONDARY OUTCOMES:
Safety: to evaluate the overall safety of allogeneic NSCLC DRibble vaccine alone or in combination with either imiquimod or GM-CSF | 43 weeks
  To evaluate the overall safety of allogeneic NSCLC DRibble vaccine alone or in combination with either imiquimod or GM-CSF, as adjuvant treatment for definitively-treated patients with Stage IIIA or B NSCLC. During the treatment period, patients will be seen in clinic 13 times over a 22-week period; performance status and side-effects will be evaluated at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, Doctor, Study Chair — The second hospital affiliated to zhejiang university school of medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xue M, Fan F, Ding L, Liu J, Su S, Yin P, Cao M, Zhao W, Hu HM, Wang L. An autophagosome-based therapeutic vaccine for HBV infection: a preclinical evaluation. J Transl Med. 2014 Dec 20;12:361. doi: 10.1186/s12967-014-0361-4. PMID 25526800
- [Background] Zhou M, Li W, Wen Z, Sheng Y, Ren H, Dong H, Cao M, Hu HM, Wang LX. Macrophages enhance tumor-derived autophagosomes (DRibbles)-induced B cells activation by TLR4/MyD88 and CD40/CD40L. Exp Cell Res. 2015 Feb 15;331(2):320-30. doi: 10.1016/j.yexcr.2014.10.015. Epub 2014 Oct 24. PMID 25447440
- [Background] Ren H, Zhao S, Li W, Dong H, Zhou M, Cao M, Hu HM, Wang LX. Therapeutic antitumor efficacy of B cells loaded with tumor-derived autophagasomes vaccine (DRibbles). J Immunother. 2014 Oct;37(8):383-93. doi: 10.1097/CJI.0000000000000051. PMID 25198526
- [Background] Ye W, Xing Y, Paustian C, van de Ven R, Moudgil T, Hilton TL, Fox BA, Urba WJ, Zhao W, Hu HM. Cross-presentation of viral antigens in dribbles leads to efficient activation of virus-specific human memory T cells. J Transl Med. 2014 Apr 16;12:100. doi: 10.1186/1479-5876-12-100. PMID 24735498